CLINICAL TRIAL: NCT04350879
Title: Evaluation of Knowledge About Contraception and Pregnancy Planning Among Type 1 and Type 2 Diabetes Women
Brief Title: Diabetes Mellitus and Pregnancy : Knowledge Assessment
Acronym: DMPKA
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20041
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; pregnancy; contraception
MeSH Terms: conditions — Diabetes Mellitus | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients: Women between 18 and 40 years old with type 1 and type 2 diabetes
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — Data record

SUMMARY:
Diabetes, a chronic and frequent disease, is a risk factor of pregnancy complications such as preeclampsia, congenital malformations and macrosomia.

Preconception care is all methods to assess the best prognostic for a diabetic pregnancy. Among these methods, contraception is very important to plan the pregnancy on a chosen moment.

The content of the preconception care is well established. However, information of diabetic women concerning contraception and giabetic pregnancy has been little studied.

DETAILED DESCRIPTION:
The aim of the study is to describe the knowledge of the patients with diabetes concerning contraception and pregnancy planning.

ELIGIBILITY:
inclusion criteria :

* Patients Aged between 18 and 40 years old
* With type 1 or type 2 diabetes mellitus
* Consulting in the department of diabetology in Reims and Charleville Mezieres hospitals
* Accepting to participate in the study

exclusion criteria :

* Patients With secondary diabetes (endocrine, pancreatic or genetical origin)
* With postmenopausal status
* Without capacity to have a pregnancy (uterine aplasia, hysterectomy)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 18 and 40 years old, consulting in diabetology department of Reims Universitary Hospital and Charleville Mézières General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Risk of unplanned pregnancy | Day 0
  Knowledge concerning the risk of unplanned pregnancy in diabete women

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Derived] Feutry L, Barbe C, Marquet-Dupont A, Fevre A, Lukas-Croisier C, Vitellius G, Delemer B, Barraud S. Contraception use and knowledge related to pregnancy in diabetic women. Ann Endocrinol (Paris). 2022 Apr;83(2):88-94. doi: 10.1016/j.ando.2022.01.007. Epub 2022 Feb 7. PMID 35143750